CLINICAL TRIAL: NCT07092033
Title: Assessment of Customized Bimodal Stimulation for Tinnitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00024155
Record Dates: First submitted 2025-07-10; First posted 2025-07-29 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Customized Bimodal Stimulation (Experimental): The study consists of one device per participant and is completed at home by the participant. Participants will be asked that bimodal stimulation is completed for one hour per day, in two 30-minute sessions every day, for the 12-week period.
  Eligible participants who consent to the study will be trained to use the device at ENROLLMENT. The 12-weeks of stimulation will consist of synchronized bimodal stimulation in which the participants' dominant tinnitus frequency will be removed from the stimulation setting via a programmed notched filter setting. A FINAL visit will be scheduled approximately 12-weeks from ENROLLMENT. Participants will be required to return their device at this visit.
  Interventions: Device: Bimodal Neuromodulation

INTERVENTIONS:
Device: Bimodal Neuromodulation — The device is a non-invasive stimulation device that consists of a controller that connects to headphones for sound delivery to the ears and connects to a mouth component that provides gentle electrical stimulation to the tongue surface. The sound is currently configured according to a tinnitus person's audiogram (i.e., hearing threshold profile for different sound frequencies) during device fitting. Individuals are recommended to use the device for 60 minutes daily (two 30-minute sessions consecutively or at different times of the day) for at least 12 weeks.

SUMMARY:
The research objective of the proposed usability study is to assess the compliance and acceptance/satisfaction of using a bimodal stimulation device with the modification of the sound stimulus to the participant's tinnitus pitch. In particular, the sound stimulus will not contain the pitch of the tinnitus, which may increase comfort and usability with the device since it will be customized to their tinnitus. Furthermore, virtual follow-up assessments and/or phone calls will be performed, thus significantly reducing the burden and personnel requirements for in-person visits as originally performed with the current clinic process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over at time of consent
* Ability to read and understand English
* Willing and able to provide and understand informed consent
* Willing to commit to the full duration of the investigation
* Subjective tinnitus
* Tinnitus duration of greater than or equal to 3 months and less than or equal to 20 years at time of consent
* Baseline Tinnitus Handicap Inventory (THI) score from 38 to 100
* Access to reliable internet connection and device to complete virtual video visits and electronic surveys
* Tonal tinnitus that can be matched

Exclusion Criteria:

* Subjective tinnitus, where pulsatility is the dominant feature
* Objective tinnitus
* Middle ear pathology in either ear including documented/known conductive hearing loss >= 20 dB at three adjacent frequencies or if a diagnosis of a tympanic membrane perforation or other middle ear pathology has been rendered, if there is an indwelling pressure equalization tube by patient report, or if middle ear surgery has been performed.
* Began wearing hearing aids within the past 3 months
* Hearing loss of greater than 80 dB HL in any test frequency in the set {2k,3k,4k,6k,8k} Hz or greater than 40 dB HL in the set {250,500,1k} Hz either unilaterally or bilaterally
* Health care provider has rendered a diagnosis of Meniere's disease or other disorder with fluctuating hearing loss
* A diagnosis of hyperacusis, misophonia or hypersensitivity to loud noises has been rendered
* History of auditory hallucinations
* Tumor on the hearing or balance nervous systems
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* Initiated new prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for a list of medical treatments.
* Ceased prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for a list of medical treatments.
* Changed dosage of prescription medications in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for a list of medical treatments.
* Any use of benzodiazepines or sedative hypnotics (either regularly or on demand)
* Neurological condition that may lead to seizures or loss of consciousness (e.g., epilepsy)
* Participant with a pacemaker or other electro-active implanted device
* Participant previously diagnosed with psychosis or schizophrenia
* Participants diagnosed with Burning Mouth Syndrome
* A diagnosis of bothersome temporomandibular joint disorder (TMJ) has been rendered
* Previous involvement in a clinical investigation for tinnitus treatment within the previous 3 months or had an implantable or surgical intervention for tinnitus
* Inability to physically or comprehensively use the device
* Oral piercings that cannot or will not be removed
* Pregnancy per patient report
* Prisoner
* Principal Investigator (PI) does not deem the candidate to be suitable for the investigation for other reasons not listed above. Rationale must be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Compliance rate after 12 weeks of bimodal stimulation | From enrollment visit to end of bimodal stimulation at 12 weeks
  Measure compliance rate in terms of the amount of time using the bimodal stimulation device over a 12 week period and demonstrate a similar rate to previous published results.

SECONDARY OUTCOMES:
Satisfaction rate after 12 weeks of bimodal stimulation | From enrollment visit to end of bimodal stimulation at 12 weeks
  Measure satisfaction rate in terms of two satisfaction questions after 12 weeks of bimodal stimulation and to demonstrate a similar rate to previous published results.

OTHER OUTCOMES:
Impact of the stimulation device on tinnitus symptoms after 12 weeks of bimodal stimulation | From enrollment visit to end of bimodal stimulation at 12 weeks
  Tinnitus Handicap Inventory (THI). The THI total scores ranges from 0 to 100, with higher scores reflecting greater severity of tinnitus handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Feng, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - PWB, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No